CLINICAL TRIAL: NCT03747432
Title: Comparison of Procedural Sedation With Propofol and Dexmedetomidine During Transcatheter Aortic Valve Implantation Using the Transfemoral Approach: Randomized Double Blind Prospective Study
Brief Title: Comparison of Procedural Sedation With Propofol and Dexmedetomidine During Transcatheter Aortic Valve Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Pia Vovk, Doctor of Medicine, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UMCLJTAVR
Record Dates: First submitted 2018-11-03; First posted 2018-11-20 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Transcatheter Aortic Valve Replacement; Procedural Sedation
Keywords: Transcatheter Aortic Valve Replacement; Procedural Sedation; Propofol; Dexmedetomidine
MeSH Terms: interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol (Experimental): Procedural sedation with propofol during the TAVR procedure (anticipated around 2 hours), dosage: 0,5-2,5 mg/kg/h for appropriate level of sedation - Ramsay sedation score 3-4)
  Interventions: Drug: Propofol
- Dexmedetomidine (Experimental): Procedural sedation with dexmedetomidine during the TAVR procedure (anticipated around 2 hours), dosage: bolus of 0,5 mcg/kg during 10 minutes, then continuous infusion of 0,2-1 mcg/kg/h for appropriate level of sedation - Ramsay sedation score 3-4)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — Procedural sedation during TAVR procedure using propofol
  Arms: Propofol
Drug: Dexmedetomidine — Procedural sedation during TAVR procedure using dexmedetomidine
  Arms: Dexmedetomidine

SUMMARY:
Aortic valve stenosis is the most common valvular heart disease in the developed world, affecting 3,9% of population over 70 years of age. If untreated it carries a poor prognosis, leading to heart failure and death in 2 years after first symptom presentation. Treatment of choice for severe aortic stenosis is surgical aortic valve replacement. A new treatment option for severe aortic stenosis emerged in the last decade - Transcatheter Aortic Valve Replacement (TAVR). This minimally invasive method was formerly reserved for high risk patients deemed unfit for surgical aortic valve replacement. Increasing use throughout the developed world and recent studies have established TAVR as a safe and viable treatment option also for intermediate-risk patients. TAVR not only enables a less aggressive surgical approach, but also a less invasive type of anaesthesia. Anaesthesiologists are trying to modify the type of anaesthesia in the way of minimally invasive approach, aiming to improve the overall outcome.

TAVR can be performed under general anaesthesia or procedural sedation (PS). From the start, TAVR was performed solely under general anaesthesia. Over time the procedure became routine and the anaesthesiologists started to commonly decide for PS. Many US and European retrospective studies have established PS to be a safe and compelling method of anaesthetic care for TAVR procedures with a favorable perioperative course, less complications, shorter intensive care unit and in-hospital stay and lower early mortality, when performed by an experienced anaesthesia team. There are many anaesthesia agents currently accepted for PS in everyday anaesthesia practice. Presently, reliable data from studies comparing different agents for PS for TAVR procedures is scarce. Most of it comes from retrospective nonrandomized trials. Propofol is a popular anaesthetic agent for PS. According to current studies, it is a safe anaesthetic agent with favorable pharmacokinetic and pharmacodynamic profiles with quite low incidence of side effects. In recent years, dexmedetomidine has been commonly used for PS having analgesic properties inclusive of its anaesthetic properties. In addition, dexmedetomidine is associated with a lesser degree of respiratory depression as to other anaesthetic agents. Patient comfort is also believed to be improved with dexmedetomidine. Studies comparing outcomes of PS with propofol versus dexmedetomidine for different non-cardiac and interventional procedures showed benefits of dexmedetomidine, owing to its analgesic properties and preferable respiratory parameters.

The aim of this study is to compare the outcome of patients undergoing TAVR under PS with dexmedetomidine against those undergoing TAVR under PS with propofol. With the results the investigators aim to aid in defining the optimal anaesthetic agent for PS for TAVR and possibly other interventional cardiology procedures.

ELIGIBILITY:
Inclusion Criteria:

* Admission to University Medical Centre Ljubljana cardiology ward for TAVR using transfemoral approach
* Voluntary agreement to participate in the study
* Aged over 18 years

Exclusion Criteria:

* Disagreement to participate in the study
* Unable to voluntarily agree to participate in the study
* Unable to participate in Mini-Mental State Examination
* History of alcohol abuse
* Diagnosed progressive dementia
* History of cerebrovascular insult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Effect of procedural sedation with propofol or dexmedetomidine on cognitive function of patients | 3 days
  The investigators will perform cognitive function testing (Mini-Mental State Examination Test) one day before the procedure (baseline result) and 48 hours after the procedure (assesing change from baseline result)
Effect of procedural sedation with propofol or dexmedetomidine on appearance of postoperative delirium | 84 hours
  The investigators will perform CAM-ICU delirium assesment method every 12 hours for 84 hours after the procedure, assesing appearance of postoperative delirium in the first 84 hours after the procedure

OTHER OUTCOMES:
Length of intensive care unit stay | 30 days after the TAVR procedure
Duration of in-hospital stay | 30 days after the TAVR procedure

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided